CLINICAL TRIAL: NCT05471362
Title: Barriers of Immediate Postpartum Intrauterine Device Uptake in Assiut Public Hospitals
Brief Title: Barriers of Immediate Postpartum Intrauterine Device Uptake
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mireille Maged Emile Hanna, Demonstrator at the Public Health Department, Assiut University
Other Study IDs: Barriers of postpartum IUD
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: IUD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases women who used IUD: Cases: women who had immediate Copper IUD inserted since October 2021 at the 4 public hospitals
  Interventions: Device: Postpartum IUD
- Control women who didn't use IUD: Controls: women who gave birth at the same hospitals and not using the immediate Copper IUD

INTERVENTIONS:
Device: Postpartum IUD — Postpartum IUD prevents pregnancy and short inter-pregnancy interval and allow spacing and family regulation
  Groups: Cases women who used IUD

SUMMARY:
increase immediate postpartum intrauterine device uptake and support family planning programs to overcome barriers and increase contraception prevalence rate in Egypt determine client related barriers of immediate postpartum intrauterine device uptake in Assiut Hospitals (Demand side) identify provider related barriers of immediate postpartum intrauterine device uptake in Assiut Hospitals (Supply side) describe method related barriers perceived by women

DETAILED DESCRIPTION:
Population increase in Egypt is a major problem with the fertility rate 3.5 children per woman the postpartum period starts after the birth of the placenta and lasts for 6-8weeks after delivery Women resume sexual activity 1 to 2 months after delivery, with 45-day average till return of ovulation. women returning for intrauterine device insertion 6-8 weeks are at risk of unintended pregnancy Insertion of postpartum intrauterine device is immediate or interval. immediate Postpartum intrauterine device inserted from the placental delivery time (within 10 minutes), or within first 48 hours, it can be done after vaginal or caesarean.

Postpartum intrauterine device can improve mothers' health by reducing difficulties from closely spaced pregnancies Immediate postpartum intrauterine device uptake is low in most developing countries and Egypt due to several barriers

* Health facility: provider knowledge, attitude, lack of training, counseling, privacy, shortage of supply of intrauterine device,poor quality of service, bad experience with the facility
* Community: as Sociodemographic (desire more children), cultural norms, husband opposition, and religious beliefs , fear of side effects., Cognitive (didn't hear about family planning in past 6 months), reproductive (long interval between intercourse), medical (requiring checkups) physical (distance of clinic) The rational is postpartum women are motivated to avoid pregnancy, 90% of women deliver in hospitals, they are in facilities with skilled physicians who can offer contraception. Immediate postpartum intrauterine device is cost-effective and efficient Assiut implemented a program training physicians on immediate Postpartum intrauterine device insertion in 2021.

This study will support the newly implemented program to overcome barriers from demand and supply sides and direct the program to future activity.

ELIGIBILITY:
Inclusion Criteria:

Women who gave birth via elective Cesarian Section at 4 public hospitals in Assiut city from October 2021:

* woman who gave birth via elective c-section at Women Health hospital of Assiut University from October 2021
* women who gave birth via elective c-section at Assiut General Hospital from October 2021
* women who gave birth at via elective c-section El-Eman El-Arbaeen from October 2021
* women who gave birth at via elective c-section El-Mabarra from October 2021

Exclusion Criteria:

* Women who delivered by vaginal delivery
* Women who delivered by emergency c-section
* women who has anomalies in the uterus

Ages: 16 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women delivering via C-Section
Study Population: Women aged from 16 to 50 who are pregnant and delivering in Assiut public hospitals via c-section
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Identifying the different barriers of uptake of immediate Postpartum copper Intrauterine device on the demand side; barriers to immediate postpartum uptake of the intrauterine device as perceived by the clients | Baseline
  Determining client related barriers of uptake of immediate postpartum copper intrauterine device in Assiut public Hospitals (Demand side) and identifying the most common barriers wether it is Cognitive; if she ever heard about Immediate postpartum intrauterine device, source of information and when was she informed about the method (during antenatal care or Delivery) and her knowledge about Immediate postpartum intrauterine device or wether it is Cultural & family factors; fertility preferences of couple, husband's or family disapproval of using contraception, fear of use due to myths and misconception, cultural preference of pregnancy in young age and the belief that untraditional contraception harm the health
Identifying the different barriers of uptake of immediate Postpartum copper Intrauterine device on the supply side; barriers as perceived by the physicians and nurses and other barriers related to the facility | Baseline
  Identifying the barriers of uptake of immediate Postpartum copper Intrauterine device on the supply side; barriers to immediate postpartum uptake of the intrauterine device as perceived by the physicians and nurses and in the facility in Assiut public hospitals such as provider personal preference, negative attitude of the hospital staff towards immediate postpartum intrauterine device, Perceived poor quality of care in the facility, previous personal or a relatives' bad experience with the facility, shortage of stock on the supply of intrauterine device in delivery settings, bad providers attitude towards pregnant women, lack of access to Postpartum intrauterine device during delivery and cost of the IUD
Identifying the method related barriers to immediate postpartum uptake of the intrauterine device as perceived by women in Assiut public hospitals | Baseline
  Describing method related barriers perceived by women such as fear of side effects, tried it before and failed, used it before and caused bleeding or pain, want the best available method, wants to try other methods, already uses a certain method and doesn't wish to change and attitude towards postpartum intrauterine device

CONTACTS AND LOCATIONS:
Overall Officials: Omaima El Gibaly, PhD, Study Director — Assiut University

REFERENCES:
- [Background] Ganatra B, Faundes A. Role of birth spacing, family planning services, safe abortion services and post-abortion care in reducing maternal mortality. Best Pract Res Clin Obstet Gynaecol. 2016 Oct;36:145-155. doi: 10.1016/j.bpobgyn.2016.07.008. Epub 2016 Aug 3. PMID 27640082
- [Background] Holden EC, Lai E, Morelli SS, Alderson D, Schulkin J, Castleberry NM, McGovern PG. Ongoing barriers to immediate postpartum long-acting reversible contraception: a physician survey. Contracept Reprod Med. 2018 Nov 8;3:23. doi: 10.1186/s40834-018-0078-5. eCollection 2018. PMID 30455978
- [Background] Eltomy EM, Saboula NE, Hussein AA. Barriers affecting utilization of family planning services among rural Egyptian women. East Mediterr Health J. 2013 May;19(5):400-8. PMID 24617117
- [Background] Divakar H, Bhardwaj A, Purandare CN, Sequeira T, Sanghvi P. Critical Factors Influencing the Acceptability of Post-placental Insertion of Intrauterine Contraceptive Device: A Study in Six Public/Private Institutes in India. J Obstet Gynaecol India. 2019 Aug;69(4):344-349. doi: 10.1007/s13224-019-01221-7. Epub 2019 May 10. PMID 31391742
- [Derived] Hanna MM, El Gibaly O, Fathalla MMF, Mohammed HM. Exploring barriers and facilitators to immediate postpartum intrauterine device uptake within the strengthening Egypt family planning program: a case-control study. BMC Health Serv Res. 2025 Aug 14;25(1):1081. doi: 10.1186/s12913-025-13306-3. PMID 40813660